CLINICAL TRIAL: NCT03966534
Title: A Randomized Controlled Study of Blood Test Draw Order to Reduce Blood Culture Contamination
Brief Title: Blood Test Order and Culture Contamination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0177-18-SZMC
Record Dates: First submitted 2019-05-21; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2018-09

CONDITIONS: Blood Culture Contamination

STUDY DESIGN:
Intervention Model Description: Prospective partially blinded randomized study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Blood culture obtained as first test after venipuncture and prior to biochemistry test
- Diversion Group (Experimental): Biochemistry test obtained as first test after venepuncture and prior to blood culture
  Interventions: Other: Blood diversion

INTERVENTIONS:
Other: Blood diversion — Diversion of initial blood obtained at venipuncture to biochemistry tube in order to try and reduce incidence of blood culture contamination
  Arms: Diversion Group

SUMMARY:
A randomized partially controlled study to examine the effect of blood diversion into a heparin lithium tube on the incidence of blood culture contamination.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Presence in Emergency Room during extended office hours (0800-2000 on weekdays(
* Clinical requirement for Blood culture and biochemistry tests from venepuncture

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Blood culture contamination | up to 7 days from obtaining blood culture
  Growth of bacteria defined as blood culture contaminants (for example coagulase negative staphylococci in one bottle only).

SECONDARY OUTCOMES:
Patient length of stay | up to 3 months from arrival
  Length of stay from arrival at Emergency room until discharge in hours

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zimmerman FS, Karameh H, Ben-Chetrit E, Zalut T, Assous M, Levin PD. Modification of Blood Test Draw Order to Reduce Blood Culture Contamination: A Randomized Clinical Trial. Clin Infect Dis. 2020 Aug 22;71(5):1215-1220. doi: 10.1093/cid/ciz971. PMID 31570942